CLINICAL TRIAL: NCT06834373
Title: Phase 2 Study of Golcadomide With Rituximab as a Bridging Therapy Prior to CAR-T for Patients With Relapsed or Primary Refractory Aggressive B-Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Golcadomide and Rituximab as Bridging Therapy for Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphoma Before CAR T-cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230813; NCI-2025-01094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-005122 (Other: Mayo Clinic Institutional Review Board); MC230813 (Other: Mayo Clinic)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Large B-Cell Lymphoma With IRF4 Rearrangement; Recurrent Aggressive B-Cell Non-Hodgkin Lymphoma; Recurrent ALK-Positive Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Recurrent Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; Recurrent Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Grade 3b Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 Rearrangements; Recurrent High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent Intravascular Large B-Cell Lymphoma; Recurrent Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Recurrent Primary Mediastinal Large B-Cell Lymphoma; Recurrent T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Refractory Aggressive B-Cell Non-Hodgkin Lymphoma; Refractory ALK-Positive Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Refractory Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; Refractory Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 Rearrangements; Refractory High Grade B-Cell Lymphoma, Not Otherwise Specified; Refractory Intravascular Large B-Cell Lymphoma; Refractory Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Refractory Primary Mediastinal Large B-Cell Lymphoma; Refractory T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; Biopsy; Immunotherapy, Adoptive; Leukapheresis; Magnetic Resonance Spectroscopy; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (golcadomide, rituximab) (Experimental): Patients receive golcadomide PO QD on days 1-14 of each cycle and rituximab IV on days 1, 8, 15 and 22 of cycle 1 and then on day 1 of all subsequent cycles. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  ELIGIBLE FOR CAR-T: After 2 cycles, patients undergo leukapheresis and may receive 1-2 additional cycles of golcadomide and rituximab prior to undergoing standard of care CAR-T therapy.
  INELIGIBLE FOR CAR-T: After 2 cycles, patients receive golcadomide PO QD on days 1-14 of each cycle and rituximab IV on day 1 of each cycle. Cycles repeat every 28 days for up to 10 additional cycles of golcadomide (cycles 3-12) and up to 3 additional cycles of rituximab (cycles 3-5) in the absence of disease progression or unacceptable toxicity.
  Patients also undergo blood sample collection and PET/CT or CT throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Biological: Chimeric Antigen Receptor T-Cell Therapy; Procedure: Computed Tomography; Drug: Golcadomide; Procedure: Leukapheresis; Procedure: Positron Emission Tomography; Biological: Rituximab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Biological: Chimeric Antigen Receptor T-Cell Therapy — Undergo standard of care CAR-T therapy
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Golcadomide — Given PO
  Other Names: BMS 986369; BMS-986369; BMS986369; CC -99282; CC 99282; CC99282; CelMod CC-99282; Cereblon E3 Ubiquitin Ligase Modulating Agent CC-99282; Cereblon E3 Ubiquitin Ligase Modulating Drug CC-99282; Cereblon Modulator CC-99282
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase II trial tests the effectiveness of golcadomide and rituximab as bridging treatment before chimeric antigen receptor (CAR) T-cell therapy in patients with aggressive B-cell non-Hodgkin lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Patients that are able to receive CAR T-cell therapy have a potential for cure, however, many will not be qualified to receive therapy due to relapse. Bridging therapy is therapy intended to transition a patient from one therapy or medication to another or maintain their health or status until they are a candidate for a therapy or have decided on a therapy. Golcadomide may help block the formation, growth or spread of cancer cells. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving golcadomide and rituximab as bridging therapy before CAR T-cell therapy may kill more tumor cells and may improve the chance of proceeding to CAR T-cell therapy in patients with relapsed or refractory aggressive B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate efficacy as measured by the disease control rate (complete metabolic response [CMR], partial metabolic response [PMR], and no metabolic response [NMR]) by Lugano 2014 positron emission tomography (PET)-computed tomography (CT) based assessment after 2 cycles of therapy.

SECONDARY OBJECTIVES:

I. To further evaluate clinical efficacy as measured by overall response rate (ORR), complete response (CMR) rate, disease control rate by Lugano PET-CT based criteria.

II. To evaluate the safety and tolerability of golcadomide + rituximab combination therapy as measured by the incidence and severity of treatment related adverse events (TRAE).

III. To evaluate efficacy as a bridging therapy as measured by the number of patients proceeding to CAR-T and response to CAR-T.

IV. To evaluate duration of response, progression-free survival, and overall survival.

EXPLORATORY OBJECTIVES:

I. Improvement of symptoms (compressive, pain, B symptoms [fever, night sweats, weight loss]) associated with the disease as determined by the investigator.

II. To evaluate the diversity of CAR-T products received in patients proceeding to CAR-T.

OUTLINE:

Patients receive golcadomide orally (PO) once daily (QD) on days 1-14 of each cycle and rituximab intravenously (IV) on days 1, 8, 15 and 22 of cycle 1 and then on day 1 of all subsequent cycles. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBLE FOR CAR-T: After 2 cycles, patients undergo leukapheresis and may receive 1-2 additional cycles of golcadomide and rituximab prior to undergoing standard of care CAR-T therapy.

INELIGIBLE FOR CAR-T: After 2 cycles, patients receive golcadomide PO QD on days 1-14 of each cycle and rituximab IV on day 1 of each cycle. Cycles repeat every 28 days for up to 10 additional cycles of golcadomide (cycles 3-12) and up to 3 additional cycles of rituximab (cycles 3-5) in the absence of disease progression or unacceptable toxicity.

Patients also undergo blood sample collection and PET/CT or CT throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy as clinically indicated.

After completion of study treatment, patients are followed up at 28 days. CAR-T ineligible patients are followed up every 3 months until progression or subsequent treatment, then every 6 months for up to 2 years. CAR-T eligible patients are followed up at 180 days after CAR-T then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed pathology diagnosis according to 2016 World Health Organization (WHO) classification including patients with diseases listed below with relapsed, progressive and/or refractory disease (Cheson et al. 2014) following treatment with one or two prior lines of standard therapy, no more than two lines of therapy are permitted:

  * Diffuse large B-cell lymphoma not otherwise specified (NOS) including:

    * Transformed lymphoma
    * Germinal center B-cell type
    * Activated B-cell type
  * High-grade B-cell lymphoma (HGBCL), NOS
  * High grade B-cell lymphoma with MYC and BCL2 translocation
  * Primary mediastinal (thymic) large B-cell lymphoma
  * Grade 3B follicular lymphoma
  * T-cell/histiocyte-rich large B-cell lymphoma
  * Large B-cell lymphoma with IRF4 rearrangement
  * Primary cutaneous diffuse large B-cell lymphoma (DLBCL), leg type
  * Epstein-Barr virus (EBV) positive DLBCL, NOS
  * DLBCL associated with chronic inflammation
  * Intravascular large B-cell lymphoma
  * ALK positive large B-cell lymphoma
  * NOTE: Richters transformation patients are excluded
* Measurable disease by PET-CT with at least one lymph node or other type of lesion that has a size > 1.5 cm in the transverse diameter, as defined by Lugano classification

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible
* Patient is potentially eligible for CAR-T therapy as determined by treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Hemoglobin > 7.0 g/dL (obtained ≤ 14 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1000/mcL (obtained ≤ 14 days prior to registration); growth factor support allowed at physician discretion
* Platelet count ≥ 75,000/mcL (obtained ≤ 14 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 14 days prior to registration); if total bilirubin is > 1.5 ULN, direct bilirubin must be normal
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN (≤ 5 x ULN if there is evidence of parenchymal liver involvement with lymphoma) (obtained ≤ 14 days prior to registration)
* Calculated creatinine clearance ≥ 45 ml/min using the Cockcroft-Gault formula (obtained ≤ 14 days prior to registration)
* Have 2 negative pregnancy tests as verified by the investigator prior to starting CC-99282:

  * A negative serum pregnancy test (sensitivity of at least 25 mIU/mL) at screening (between 10 to 14 days prior to cycle 1 day 1)
  * A negative serum or urine pregnancy test (investigator's discretion) within 24 hours prior to cycle 1 day 1 of study treatment
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Subjects must agree not to donate blood while receiving golcadomide, during dose interruptions and for ≥ 28 days following the last dose of golcadomide

Exclusion Criteria:

* Any of the following because this study involves an investigational agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
* Persons of childbearing potential (and persons able to father a child) who are unwilling to employ adequate contraception

  * Persons of childbearing potential (PCBP) unwilling to use two reliable forms of contraception simultaneously or to practice complete abstinence (true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g., calendar, ovulation, symptothermal or postovulation methods] and withdrawal are not acceptable methods of contraception) from heterosexual contact during the following time periods related to this study:
  * For ≥ 28 days before starting treatment, during treatment and dose interruptions, and for ≥ 28 days after the last dose of golcadomide
  * Examples of highly effective methods of contraception:

    * Intrauterine device (IUD)
    * Hormonal (birth control pills, injections, implants, levonorgestrel-releasing intrauterine system [IUS], medroxyprogesterone acetate depot injections, ovulation inhibitory
    * Progesterone-only pills [e.g., desogestrel])
    * Tubal ligation
    * Partner's vasectomy
  * Examples of additional effective methods:

    * Male condom
    * Diaphragm
    * Cervical cap
  * Persons who can father a child unwilling to practice complete abstinence (true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g., calendar, ovulation, symptothermal or post-ovulation methods] and withdrawal are not acceptable methods of contraception.) or unwilling to use a condom during sexual contact with a pregnant person or a PCBP during treatment and dose interruptions, and for > 28 days following the last dose of golcadomide, even if they have undergone a successful vasectomy
  * Persons who can father a child and are unwilling to refrain from donating semen or sperm while receiving golcadomide, during dose interruptions, or for ≥ 28 days following the last dose of golcadomide
* Life expectancy < 3 months
* Any of the following prior therapies:

  * Any prior CAR-T or other T-cell targeting treatment (approved or investigational) ≤ 4 weeks prior to registration
  * Any prior systemic anti-cancer treatment (approved or investigational) ≤ 5 half-lives or 4 weeks prior to registration, whichever is shorter

    * Exception: Monoclonal and bispecific antibodies is acceptable
  * Prior therapy with golcadomide ≤ 4 weeks prior to registration
  * Prior autologous stem cell transplantation (SCT) ≤ 3 months prior to registration. If subject had autologous SCT > 3 months prior to the start of registration, any treatment-related toxicity is unresolved (grade > 1)
  * Major surgery ≤ 3 weeks prior to registration
  * Chemotherapy ≤ 2 weeks prior to registration
  * Concomitant radiation therapy; local palliative radiotherapy is permitted
* Co-morbid systemic illnesses or other severe concurrent disease or cancer which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Impaired cardiac function or clinically significant cardiac diseases including, but not limited to:

  * Symptomatic congestive heart failure
  * History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy (such as interstitial lung disease or chronic obstructive pulmonary disease [COPD])
  * Any other conditions that would limit compliance with study requirements
* Subject had prior allogeneic SCT with either standard or reduced intensity conditioning ≤ 6 months prior to registration. If subject had prior allogeneic SCT > 6 months prior to registration, any treatment-related toxicity is unresolved (grade >1)
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy, as there is currently no safety data in HIV positive patients
* Subject has known chronic active hepatitis B or C virus (HBV/HCV) infection

  * Exception: Patients with HBV and an undetectable viral load who are on suppressive therapy and/or those with HCV and an undetectable viral load are allowed
* Concurrent administration of strong or moderate CYP3A4/5 inhibitors and inducers within 14 days or 5 half-lives, whichever is longer before the study treatment administration
* Receiving any other investigational agent which would be considered as a treatment for lymphoma.

  * Exception: Corticosteroids are allowed
* Active second malignancy requiring treatment that would interfere with the assessment of the response of the primary cancer or interpretation of the safety of this protocol therapy
* History of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia. Patients with a history of deep vein thrombosis (DVT)/pulmonary embolism (PE) or thrombophilia may still participate if they are willing to be on full anticoagulation during treatment. Full anticoagulation is defined as Warfarin, factor X inhibitors, or low molecular weight heparin at therapeutic doses. The rationale for this requirement is that golcadomide therapy is associated with an increased risk of thrombosis. Patients with no history of DVT/PE or thrombophilia are not required to take anticoagulation and/or anti-platelet prophylaxis

  * NOTE: If a patient develops a thrombotic event, they must be able and willing to receive anticoagulation therapy with aspirin 81-325 mg daily prophylaxis, low molecular weight heparin, factor X inhibitors or Warfarin. This is due to an increased risk of thrombosis in patients treated with golcadomide without prophylaxis
* Live COVID-19 vaccine administered ≤ 28 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Disease control | 2 cycles (cycle length = 28 days)
  Will be defined as a complete metabolic response (CMR), partial metabolic response (PMR), or no metabolic response (NMR) by Lugano 2014 PET-CT.

SECONDARY OUTCOMES:
Disease control rate | Up to 2 years
  Will be estimated by the total number of patients who achieve a CMR, PMR, or NMR by Lugano 2014 positron emission tomography (PET)/computed tomography (CT) divided by the total number of evaluable patients.
Complete response rate | Up to 2 years
  Will be assessed by the total number of patients who achieve a CMR by Lugano 2014 PET/CT.
Overall response rate | Up to 2 years
  Will be assessed by the total number of patients who achieve a CMR or PMR by Lugano 2014 PET/CT divided.
The proportion of patients proceeding to chimeric antigen receptor T-cell (CART) | Up to 2 years
  Will be assessed by the total number of patients who proceed to CART divided by the total number of evaluable patients.
Overall response rate to CART | Up to 2 years
  Will be assessed by the total number of patients who achieve a CMR or PMR by Lugano 2014 PET/CT after CART.
Duration of response | Up to 2 years
  Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CMR or PMR to first documentation of disease progression.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from registration to first documentation of disease progression (PMD or PD) or death due to any cause in the absence of documented progression
Overall survival (OS) | From registration to death due to any cause, assessed up to 2 years
  Overall survival is defined as the time from registration to death due to any cause.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE). The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration and treatment related AEs will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Tiger, MD, PhD, Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials